CLINICAL TRIAL: NCT01363479
Title: Single-dose, Multicenter, Randomized, Double-blind, Double-dummy, Parallel Group Study to Assess the Efficacy and Safety of Oral Palonosetron 0.50 mg Compared to I.V. Palonosetron 0.25 mg Administered With Dexamethasone for the Prevention of Chemotherapy-induced Nausea and Vomiting in Cancer Patients Receiving Highly Emetogenic Cisplatin-based Chemotherapy
Brief Title: An Efficacy and Safety Study of Oral and Intravenous Palonosetron for the Prevention of Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALO-10-01
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral palonosteron plus dexamethasone (Experimental): Oral palonosetron (Aloxi 0.50 mg softgel capsule) with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Interventions: Drug: Oral palonosetron; Drug: Dexamethasone
- I.V. palonosetron plus dexamethasone (Active Comparator): Intravenous palonosetron (Aloxi 0.25 mg solution for injection) with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Interventions: Drug: I.V. palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Oral palonosetron
  Arms: Oral palonosteron plus dexamethasone
Drug: I.V. palonosetron
  Arms: I.V. palonosetron plus dexamethasone
Drug: Dexamethasone

SUMMARY:
PALO-10-01 is a clinical study assessing efficacy and safety of a single oral dose of palonosetron compared to a single intravenous dose of palonosetron (Aloxi, an antiemetic drug), both given with oral dexamethasone. The objective of the study is to demonstrate that oral palonosetron 0.50 mg is as effective as (non-inferior to) palonosetron IV 0.25 mg to prevent nausea and vomiting induced by highly emetogenic cancer chemotherapy in the 0-24 hours after administration of a single cycle of highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Naïve to cytotoxic chemotherapy. Previous biological or hormonal therapy is permitted.
* Diagnosed with a malignant solid tumor and scheduled to receive first course of cytotoxic chemotherapy with cisplatin administered as a single I.V. dose of equal or more than 70 mg/m2 over 1-4 hours on study Day 1, either alone or in combination with other chemotherapeutic agents.
* If scheduled to receive combination regimens, non-cisplatin agents of moderate to high emetogenic potential are allowed and they must be administered following the cisplatin infusion and completed no more than 6 hours after the initiation of cisplatin infusion.
* If scheduled to receive chemotherapy agents of minimal to low emetogenic potential, they are to be given on Day 1 following cisplatin or on any subsequent study day.
* ECOG Performance Status of 0, 1, or 2
* Female patients of either non-childbearing potential or child-bearing potential with a commitment to use contraceptive methods throughout the clinical trial
* Hematologic and metabolic status adequate for receiving a highly emetogenic cisplatin-based regimen based on laboratory criteria (Neutrophils,Platelets, Bilirubin, Liver enzymes, Serum Creatinine or Creatinine Clearance)
* If a patient has a known hepatic or renal impairment, he/she may be enrolled in this study at the discretion of the Investigator.
* If a patient has a known history or predisposition to cardiac conduction interval abnormalities he/she may be enrolled in this study at the discretion of the Investigator.

Exclusion Criteria:

* If female, pregnant or lactating.
* Current use of illicit drugs or current evidence of alcohol abuse.
* Scheduled to receive moderately emetogenic chemotherapy (MEC) or HEC from Day 2 to Day 5 following cisplatin administration.
* Received or is scheduled to receive radiation therapy to the abdomen, or the pelvis within 1 week prior to Day 1 or between Days 1 to 5.
* Any vomiting, retching, or mild nausea within 24 hours prior to Day 1.
* Symptomatic primary or metastatic CNS malignancy.
* Active peptic ulcer disease, gastrointestinal obstruction, increased intracranial pressure, hypercalcemia, an active infection or any uncontrolled medical conditions (other than malignancy) that, in the opinion of the investigator, may confound the results of the study, represent another potential etiology for emesis and nausea (other than chemotherapy-induced nausea and vomiting, CINV) or pose unwarranted risks in administering the study drugs to the patient.
* Known hypersensitivity or contraindication to 5-HT3 receptor antagonists (e.g., palonosetron, ondansetron, granisetron, dolasetron, tropisetron, ramosetron) or dexamethasone.
* Participation in a clinical trial involving palonosetron.
* Any investigational drugs (other than those given in this study) taken within 4 weeks prior to Day 1, and/or is scheduled to receive any investigational drug during the study.
* Systemic corticosteroid therapy at any dose within 72 hours prior to Day 1. However topical and inhaled corticosteroids with a steroid dose of £ 10 mg of prednisone daily or its equivalent are permitted.
* Scheduled to receive bone marrow transplantation and/or stem cell rescue therapy.
* Any medication with known or potential antiemetic activity within 24 hours prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (9):
  - Genesis Cancer Centre, Hot Springs, Arkansas
  - Compassionate Cancer Center, Corona, California
  - Compassionate Cancer Centre Medical Group, Fountain Valley, California
  - Facey Medical Group, Mission Hills, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Wellmont Medical Associates-Oncology and Hematology, Bristol, Rhode Island
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Northern Utah Associates [Hematology/ Oncology], Ogden, Utah
- Argentina (7):
  - Centro Oncológico Integral (COI), Mar del Plata, Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Instituto Oncológico de Córdoba (IONC), Córdoba
  - Instituto Médico CER [Oncology], Quilmes
  - Sanatorio Parque, Rosario
  - Centro Medico San Roque, San Miguel de Tucumán
  - ISIS Clinica Especializada, Santa Fe
- Bulgaria (6):
  - MHAT Dr. Tota Venkova, Gabrovo
  - Specialized Hospital for Active Treatement of Oncology Diseases - Sofia District Medical Oncology Department, Sofia
  - UMHAT "Tsaritsa Yoanna - ISUL" Ltd.Medical Oncology Clinic, Sofia
  - Specialised Hospital for Active treatment on Oncology, Sofia
  - District Dispensery for Oncology Diseases with in-patient, Sofia
  - Complex Oncology Centre, Stara Zagora
- Croatia (5):
  - Klinicki bolnicki centar [Oncology], Osijek
  - KBC Rijeka, Rijeka
  - Opca bolnica Varazdin, Varaždin
  - KBC Zagreb, Zagreb
  - Klinicka bolnica [Sestre milosrdnice], Zagreb
- Germany (4):
  - Klinik und Poliklinik für Onkologie und Hämatologie Universitätsmedizin Charité Mitte, Berlin
  - OncoResearch Lerchenfeld UG, Hamburg
  - Städtisches Klinikum München, München
  - Staedtisches Krankenhaus Muenchen Neuperlach, München
- Hungary (6):
  - Semmelweis Egyetem Kútvölgyi Klinikai Tömb, Budapest
  - Fővárosi Önkormányzat Uzsoki utcai Kórház, Budapest
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Bács-Kiskun Megyei Önkormányzat Kórháza, Szeged, Kecskemét
  - Pécsi Tudományegyetem [Onkoterápiás Intézet], Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz, Szolnok
- India (6):
  - Yashoda Super speciality Hospital, Hyderabad, Andhra Pradesh
  - Sujan Surgical Cancer Hospital and Amracvati Cancer Foundation, Pune, Maharashtra
  - Apollo Speciality Hospital, Chennai, Tamil Nadu
  - Sri Venkateshwara Hospital [Medical Oncology], Bangalore
  - Chinmaya Mission Hospital, Bangalore
  - City Cancer Centre [Surgical and Medical Oncology], Vijayawada
- Italy (4):
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Ospedale Vito Fazzi - ASL Lecce, Lecce
  - Presidio Ospedaliero "Alessandro Manzoni", Lecco
  - AO Regionale S.Carlo di Potenza, Potenza
- Poland (6):
  - Szpital Wojewodzki Zespolony, Elblag
  - Wojewodzki Szpital Specjalistyczny im. M.Kopernika, Lodz
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej - Curie, Warsaw
  - NZOZ Magodent - Centrum Medczyne Ostrobramska, Warsaw
  - Szpital Wojewodzki w Lomzy im. Kardynala S. Wyszynskiego, Łomża
- Romania (8):
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris", Baia Mare
  - Institutul Oncologic "Prof. Dr. Alex. Trestioreanu", Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj (Oncologie Medicala), Cluj-Napoca
  - Centrul de Oncologie Euroclinic, Iași
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu [Oncologie], Sibiu
  - Oncomed SRL, Timișoara
- Russia (11):
  - GUZ Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk
  - GOU VPO Krasnoyarsk State Medical University n.a. prof. V.F., Krasnoyarsk
  - GUZ Lipetsk Regional Oncology Dispensary [General Oncology], Lipetsk
  - GUZ Regional Oncology Dispensary #2, Magnitogorsk
  - RAMN - Russian Cancer Research Center, Moscow
  - Russian Oncology Research Center n.a. N.N. Blokhin RAMN, Moscow
  - MBUZ City Clinical Hospital #1 [Oncology], Novosibirsk
  - FGBU "Medical Radiology Scientific Center of Minzdravsotsrazvitiya RF, Obninsk
  - Ryazan State Med. Univer. n.a. I.I.Pavlov based Ryazan Regio, Ryazan
  - GUZ Leningrad Regional Oncological Dispensary, Saint Petersburg
  - St. Petersburg Clinical Oncology Dispesary, Saint Petersburg
- Ukraine (7):
  - Komunalnyi likuvalno-profilaktychnyi zaklad "Chernigivskyi, Chernihiv
  - Komunalnyi zaklad Miska bahatoprofilna klinichna likarnia #4, Dnipropetrovsk
  - Komunalno-klinichnyi likuvalno-profilaktychnyi zaklad, Donetsk
  - DU IMR AMNU [vd khemter], Kharkiv
  - Kharkivskyi oblasnyi onkologichnyi klinichnyi tsentr, Kharkiv
  - Chmelnytskyi Regional Clinical Oncology Centre [Oncology], Khmelnytskyi
  - Uzhgorod National University, Uzhhorod

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 743 patients were randomized (ITT population), 739 received study medications (oral or I.V. palonosetron plus dexamethasone, safety population), 738 received study medications (oral or I.V. palonosetron plus dexamethasone, safety population) and chemotherapy (FAS population)
Groups:
- Oral Palonosteron Plus Dexamethasone: Oral palonosetron (Aloxi 0.50 mg softgel capsule) with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Oral palonosetron
  Dexamethasone
- I.V. Palonosetron Plus Dexamethasone: Intravenous palonosetron (Aloxi 0.25 mg solution for injection) with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  I.V. palonosetron
  Dexamethasone
Period: Overall Study
Arm/Group | Oral Palonosteron Plus Dexamethasone | I.V. Palonosetron Plus Dexamethasone
Started | 371 (number of randomised patients) | 372 (number of randomised patients)
Completed | 359 | 351
Not Completed | 12 | 21

BASELINE CHARACTERISTICS:
Population: Safety population ie patients receiving either oral or IV palonosetron plus dexamethasone
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Palonosteron Plus Dexamethasone | I.V. Palonosetron Plus Dexamethasone | Total
Number analyzed (Participants) | 370 | 369 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (9.41) | 57.7 (9.92) | 57.9 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 152 | 303
  Male | 219 | 217 | 436
Race/Ethnicity, Customized [Number; unit: participants]
  White | 321 | 320 | 641
  Asian | 49 | 47 | 96
  Hispanic | 0 | 1 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication
Time Frame: 0-24 hours
Population: Full Analysis Set i.e. patients receiving study drugs and chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Oral Palonosteron Plus Dexamethasone | I.V. Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 369 | 369
percentage of responders | 89.4 [85.9 to 92.2] | 86.2 [82.3 to 89.3]
Statistical Analysis 1: Comparison: Oral Palonosteron Plus Dexamethasone vs I.V. Palonosetron Plus Dexamethasone; Test type: Non-Inferiority or Equivalence — The null hypothesis was rejected (and non inferiority of oral palonosetron 0.50 mg versus I.V. palonosetron 0.25 mg demonstrated), if the lower limit of the 2 sided 99% CI for the difference in proportion of patients with CR (risk difference) was greater (i.e., closer to zero) than 15%.Study had 90% power; Risk Difference (RD) = 3.21, 99% CI 2-sided [-2.74 to 9.17] — The risk difference and the 99% CI calculation were performed using a 2 sided stratum adjusted Cochran Mantel Haenszel (CMH) test including gender and region as strata

2. Secondary Outcome: Percentage of Patients With no Emesis
Time Frame: 0-24 hours
Population: FAS i.e. patients receiving study drugs and chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Oral Palonosteron Plus Dexamethasone | I.V. Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 369 | 369
percentage of responders | 90.2 [86.8 to 92.9] | 86.7 [82.9 to 89.8]

3. Secondary Outcome: Percentage of Patients With no Rescue Medication
Time Frame: 0-24 hours
Population: FAS i.e. patients receiving study drugs and chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Oral Palonosteron Plus Dexamethasone | I.V. Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 369 | 369
percentage of responders | 94.6 [91.8 to 96.5] | 93.2 [90.2 to 95.4]

ADVERSE EVENTS:
Time Frame: Period starting from the time of informed consent signature until 21 days post study drugs administration on Day 1.
Description: Based on the medical judgment of the investigator, all non resolved, non serious AEs beyond this date could have been followed for an additional 14 days. At the end of this additional follow up period, all unresolved AEs were documented on the eCRF as "ongoing."
Arm/Group | Oral Palonosteron Plus Dexamethasone | I.V. Palonosetron Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 36/370 | 36/369
Other Adverse Events (participants affected / at risk) | 168/370 | 171/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Palonosteron Plus Dexamethasone (N=370) | I.V. Palonosetron Plus Dexamethasone (N=369)
Anemia (Blood and lymphatic system disorders) | 1 | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Leucopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 9
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Aphagia (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 3 | 1
Chest Pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 4
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngotracheal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Palonosteron Plus Dexamethasone (N=370) | I.V. Palonosetron Plus Dexamethasone (N=369)
Neutropenia (Blood and lymphatic system disorders) | 21 | 28
Constipation (Gastrointestinal disorders) | 23 | 20
Asthenia (General disorders) | 31 | 28
Decreased appetite (Metabolism and nutrition disorders) | 21 | 11
Headache (Nervous system disorders) | 9 | 21
Investigations (Investigations) | 41 | 45
Respiratory, thoracic and mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 22 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor and investigator(s) agree that no publications discussing trials' results will occur until release of final report. Sponsor has no objections if the investigators publish study results, however the investigator is requested to contact the sponsor before publishing, to prevent premature disclosure of data and is not intended as a restrictive measure concerning results or opinions of investigators.